CLINICAL TRIAL: NCT06259747
Title: Potential Therapeutic Implications of Acutaping on Nausea and Vomiting During Pregnancy
Brief Title: Therapeutic Implications of Acutaping on Nausea and Vomiting During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Mennat Allah Hassan Mohamed Elghoul, Demonstrator at women's health department, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Acutaping for NVP
Record Dates: First submitted 2024-02-07; First posted 2024-02-14 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Nausea; Vomiting of Pregnancy
MeSH Terms: conditions — Nausea | interventions — dicyclomine, doxylamine, pyridoxine drug combination

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated into two groups; group (A) will receive acutaping in addition to traditional medical treatment (Doxylamine and Pyridoxine) while group (B) will receive traditional medical treatment(Doxylamine and Pyridoxine) only.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- acutaping and traditional medical treatment (Experimental): received acutaping in addition to traditional medical treatment (Doxylamine and Pyridoxine)
  Interventions: Other: Acutaping; Drug: Doxylamine and Pyridoxine
- traditional medical treatment only (Experimental): received traditional medical treatment only (Doxylamine and Pyridoxine
  Interventions: Drug: Doxylamine and Pyridoxine

INTERVENTIONS:
Other: Acutaping — Application of the kinesio tape on finger and forearm flexor tape after localization of the acupoints of application
  Arms: acutaping and traditional medical treatment
Drug: Doxylamine and Pyridoxine — traditional medical treatment for nausea and vomiting during pregnancy

SUMMARY:
This study will answer the following research question:

Is acutaping has therapeutic implications on symptoms of nausea and vomiting during pregnancy?

DETAILED DESCRIPTION:
Nausea and vomiting during pregnancy (NVP) are common symptoms, with prevalence rate from 50% to 90% . NVP symptoms often appear between weeks 5 and 6, peak at 8 to 9 weeks, and subside between weeks 16 and 20 .Long-term morning sickness during pregnancy increases the incidence of postpartum depression symptoms in women and severe NVP increases the chance of low birth weight .

NVP is multifactorial and the most common causes potentially including hormone imbalances, placental disorders, and genetic causes . Genetic factors, Evidence in support of a genetic predisposition to nausea and vomiting of pregnancy includes the following: (a) the concordance in frequency of nausea and vomiting of pregnancy in monozygotic twins ; (b) the finding that siblings and mothers of patients affected with nausea and vomiting of pregnancy are more likely to be affected than relatives of unaffected individuals ; (c) the variation in frequency between ethnic groups; (d) the higher frequency of nausea and vomiting of pregnancy in patients with predisposing conditions that are genetically determined such as taste sensation; and (e) the occurrence of nausea and vomiting of pregnancy in women with inherited glycoprotein hormone receptor defects.

The fundamental stimulus-a placental product, the triggering factor for nausea and vomiting of pregnancy has not been identified, although human chorionic gonadotropin and estrogens have been implicated. The principle reason for considering human chorionic gonadotropin initially was the close temporal association between peak human chorionic gonadotropin concentrations and peak nausea and vomiting of pregnancy symptoms. Conditions associated with higher human chorionic gonadotropin production are associated with nausea and vomiting of pregnancy. These include multiple gestation with hyperemesis gravidarum 4 to 5 times more common than in singletons .

Whatever the specific trigger, the emetic response is fundamentally the same: there is a marked reduction in gastric tone and motility followed by a retrograde giant contraction moving small intestinal contents into the stomach. Thereafter, contractions of the diaphragm and abdominal muscles combine with relaxation of the gastroesophageal sphincter to facilitate passage of gastrointestinal contents .

Although there are several pharmacological treatments for NVP, many medical professionals and expectant mothers prefer non-pharmacological therapy over pharmacological ones because of worry for their impact on foetal outcomes .

For years, traditional Chinese acupuncture has been promoted as a helpful antiemetic . An alternative treatment for preventing nausea and vomiting is acupressure .

Kinesio tape is an elastic therapeutic tape that is drug free and used to treat a range of musculoskeletal issues, including dysfunction, pain, and injury and a variety of other disorders .When compared to normal drugs alone, kinesio taping on the stomach area is more successful at relieving nausea and vomiting in emesis gravidarum patients .

In acutaping, acupressure/acupuncture and kinesio taping are used to treat internal and gynecological issues like nausea and vomiting during pregnancy by stimulating acupressure points with kinesio tape .

Nausea and vomiting of pregnancy is a very common disorder reported in 70-80% of all pregnant women . The extent of vomiting may be so profound that weight loss, electrolyte imbalance, and dehydration requiring hospitalisation result . Women with nausea and vomiting during pregnancy and nausea only during pregnancy had proteinuria and preeclampsia than the symptom free women .NVP also has a significant detrimental impact on quality of life (QoL) , especially affecting physical QoL and work function. This impact is evident across the spectrum of NVP, but significantly worse with more severe symptoms .

Studies have repeatedly shown that there is a high perception of teratogenic risk among pregnant and planning women regarding medication use in pregnancy , and that this is also true for NVP , which is experienced by the vast majority of pregnant women.

There are many studies using acustimulation on nausea and vomiting in pregnant women including acupressure, acupuncture, and electrical stimulation.The stimulation of this point can also be done by dry cupping and also auriculotherapy used for NVP .

There is no study about the potential therapeutic implication of acutaping on nausea and vomiting during pregnancy, so our study will be used to detect this therapeutic implication of acutaping.

ELIGIBILITY:
Inclusion Criteria:

* Woman with nausea and vomiting during pregnancy Primigravida With age ranges from 20-35years Gestational age 7-16 weeks Body mass index (BMI) less than 30 kg/m2 Not hospitalized due to hyperemesis gravidarum

Exclusion Criteria:

* Gastrointestinal disorder Diabetes Dehydration

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women
Enrollment: 27 (Actual)
Dates: Start 2023-02-03 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
pregnancy unique quantification of emesis and nausea questionnaire | Measured before treatment , after first treatment (at 4th day) and after second treatment (at 8th day )
  Frequency of nausea & vomiting and dry heaviness without vomiting Score.
  detection of frequency of nausea & vomiting and dry heaviness without vomiting , total score of frequency of nausea & vomiting and dry heaviness without vomiting (sum of replies to 1, 2, 3 questions): Mild NVP ≤ 6, Moderate NVP 7-12, severe NVP ≥ 13.
pregnancy unique quantification of emesis and nausea questionnaire | Measured before treatment , after first treatment (at 4th day) and after second treatment (at 8th day )
  Quality of life in those pregnant women Score the quality of life question is on a scale of 0-10 with: 0(worst possible), 10 (as good as you felt before pregnancy).

CONTACTS AND LOCATIONS:
Overall Officials: Eman Abdelfatah Elhosary, professor at women's health, Study Director — Women's Health Department ,Faculty Of Physical Therapy Kafr Elsheikh University; Fayiz Farouk Elshamy, professor at women's health, Study Director — Women's Health Department ,Faculty Of Physical Therapy Kafr Elsheikh University; Tamer Mahmoud Zaki, Fellow Obst. and gyna., Study Director — Obestetrics And Gynecology Depatment, Damanhour Teaching Hospital
Locations (1):
- Damanhour teaching hospital and private clinics, Kafr ash Shaykh, Egypt